## The Effect of White Light on Fatigue Levels in Patients With Gynecological Cancer: A Double Blind Randomized Trial

## 02.08.2021

## INFORMATION CONSENT FORM

Cancer-related fatigue; Resistant, subjective physical, emotional, and/or cognitive fatigue or burnout associated with cancer and cancer treatment. This condition has different severity and rates before, during and after treatment. Cancer-related fatigue occurs due to common complaints such as diseases, side effects of treatment, sleep problems, pain, nausea and vomiting. Therefore, patients should be routinely evaluated and managed according to diagnosis, treatment and disease stage. Fatigue management should include drug and non-drug interventions planned for the individual according to the period of the patient (treatment, post-treatment and last period). When the studies and guidelines are evaluated, education, counseling, physical activity, yoga, acupressure, massage, cognitive-behavioral therapy, psycho-educational therapy, meaningful supportive therapies, nutritional support, cognitive-behavioral therapy for sleep, bright white light application in the non-drug management of fatigue is located. Among these treatments, white light application, which has no side effects and has a low cost, is known to reduce fatigue by regulating the circadian rhythm. Therefore, this research was planned as a scientific research project to evaluate the effect of white light on fatigue in gynecological-oncology patients.

The study was designed in two groups and the fatigue status of the patients in the application and control groups will be evaluated, while 10,000lux white light will be applied to the patients in the application group, routine nursing interventions will be applied to the patients in the control group. Which of these groups you will be included in will be determined by the method of the table of numbers obtained on the computer. During the research, you will not be given any drug treatment or any harmful application other than the treatment planned by your doctor.

With your participation in this study, the effect of white light to be applied on fatigue management will be determined. Your name and information on the form will remain with us and will not be used for any other purpose.

| I I | Individual introduction | form contain | ing the inform | nation |
|---|---|---|---|---|
| they want me to answer in order to de | etermine the situations r | related to my | fatigue status | during |
| my illness and treatment, to answer the | he questionnaires in the | Brief Fatigue | Inventory, to | apply |
| white light if I am in the application § | group. I voluntarily acce | ept. | | |

## DATE:

Patient The relatives of the patient Researcher

(Name-Surname-Signature)